CLINICAL TRIAL: NCT05307458
Title: Evaluating the Pharmacokinetics and Patient Outcomes of Buprenorphine Microdosing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: United Health Services Hospitals, Inc. (Other)
Collaborators: Binghamton University (Other)
Responsible Party: Principal Investigator, William Eggleston, Assistant Professor, Binghamton University
Other Study IDs: 11453
Record Dates: First submitted 2022-03-17; First posted 2022-04-01 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Opioid Use Disorder; Opioid Withdrawal
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Buprenorphine Microdosing: Participants transitioning to buprenorphine from methadone using a microdosing protocol.
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Participants will receive gradually increasing doses of buprenorphine while tapering down on their methadone dose.

SUMMARY:
There are more than 2.1 million people in the United States with opioid use disorder, and according to preliminary data from the US Centers for Disease Control and Prevention opioid overdose deaths rose 36% to more than 69,000 deaths in 2020. Treatment with buprenorphine or methadone reduces overdose deaths in patients with opioid use disorder. However, most patients with opioid use disorder do not receive treatment. In addition to the rising rates of morbidity and mortality, the healthcare, social, and societal costs of the opioid epidemic are roughly one trillion dollars annually. Rapidly scalable strategies are needed to increase access to treatment and improve treatment retention.

The investigators propose a novel buprenorphine micro-dosing study to evaluate the pharmacokinetics, treatment retention, and qualitative outcomes in participants transitioning from methadone maintenance therapy to buprenorphine using a micro-dosing initiation in the outpatient setting. The proposed study will report participant pharmacokinetics, treatment retention, Clinical Opiate Withdrawal Scale (COWS) score, Treatment Satisfaction Questionnaire for Medication (TSQM) score, and other qualitative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include adults (at least 18 years of age) who have been enrolled and receiving consistent treatment in the methadone program for at least 6 months.

Exclusion Criteria:

* Participants will be excluded if they are on a methadone dose > 80 mg, have concurrent alcohol use or benzodiazepine use disorder, require opioids for a pain-related diagnosis, are a current suicide or homicide risk, have a current psychotic disorder (DSM-V) or untreated major depression, have a life-threatening or unstable medical problem, or are pregnant.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will include adults (at least 18 years of age) who have been enrolled and receiving consistent treatment in the methadone program for at least 6 months. Participants will be excluded if they are on a methadone dose > 80 mg, have concurrent alcohol use or benzodiazepine use disorder, require opioids for a pain-related diagnosis, are a current suicide or homicide risk, have a current psychotic disorder (DSM-V) or untreated major depression, have a life-threatening or unstable medical problem, or are pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid withdrawal symptoms | 14-days
  Opioid withdrawal symptoms will be measured using the clinical opiate withdrawal scale (COWS) score and subjective opiate withdrawal scale (SOWS) score.

SECONDARY OUTCOMES:
Acute Precipitated Withdrawal | 14-days
  Severe opioid withdrawal symptoms resulting in hospitalization.
Treatment retention | 6-months
  Patient retention in the buprenorphine treatment program. Defined as continued treatment with buprenorphine.
Area Under the Curve | 14-days
  Buprenorphine AUC will be measured in participants.
Peak concentration | 14-days
  Buprenorphine peak concentrations will be measured in participants.

CONTACTS AND LOCATIONS:
Locations (1):
- UHS Addiction Medicine, Binghamton, New York, United States

IPD SHARING:
Plan to Share IPD: No